CLINICAL TRIAL: NCT02024880
Title: A Randomized Single-blind Comparison of Two Embryo Transfer Catheters in Patients Undergoing in Vitro Fertilization and Embryo Transfer
Brief Title: Comparison of Two Embryo Transfer Catheters in Patients Undergoing in Vitro Fertilization and Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The ET catheters were outdated.
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKUQMHCARE002
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2020-07

CONDITIONS: Infertility
Keywords: in vitro fertilization; embryo transfer; transfer catheter
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protective catheter group (Experimental): Protective catheter group uses Guardia™ Pro Protective ET catheter from Cook.
  Interventions: Device: Protective catheter group
- Conventional catheter group (Active Comparator): Conventional catheter group uses Sydney IVF catheter from Cook.
  Interventions: Device: Conventional catheter group

INTERVENTIONS:
Device: Protective catheter group — The tip of this catheter is protected on insertion of the catheter.
  Other Names: Guardia™ Pro Protective ET catheter
  Arms: Protective catheter group
Device: Conventional catheter group — A standard embryo catheter
  Other Names: Sydney IVF catheters
  Arms: Conventional catheter group

SUMMARY:
In-vitro fertilization (IVF) treatment involves development of multiple follicles following ovarian stimulation, oocyte retrieval and embryo transfer (ET). ET is the final and most crucial step of IVF treatment.

The ET catheter has to pass through the endocervical canal to go into the uterine cavity through the internal os. The endocervical canal may be filled up with mucus or blood. Embryos trapped in the mucus or blood after the passage of the endocervical canal may not be able to implant into the endometrium. Guardia™ Pro Protective ET catheter is designed to allow the safe passage of embryos through cervical mucus and blood as its outer sheath protects the embryo through entry and then opens in petals to further advance the inner catheter and gently place the embryo.

The hypothesis of this study is that the pregnancy rate is significantly higher after ET using protective ET catheters.

DETAILED DESCRIPTION:
In-vitro fertilization (IVF) treatment involves development of multiple follicles following ovarian stimulation, oocyte retrieval and embryo transfer (ET). Despite recent advances in ovarian stimulation, the method of assisted fertilization and improved culture conditions, the implantation potential of embryos remains around 20-25% for a long time.

ET is the final and most crucial step of IVF treatment and pregnancy rates after ET may be affected by various factors. In a Cochrane meta-analysis (Derks et al., 2009), no evidence of a benefit was found for performing ET with a full bladder, the removal of cervical mucus, and flushing the endocervical canal or the endometrial cavity. No data were found on changing the woman's position, the use of a tenaculum, the performance of a dummy transfer, and embryo afterloading. Other meta-analyses demonstrate that the use of soft ET catheters (Buckett, 2008) and transabdominal ultrasound guidance (Brown et al., 2010) lead to a higher chance of clinical pregnancy when compared with the use of stiff catheters and clinical touch respectively.

The ET catheter has to pass through the endocervical canal to go into the uterine cavity through the internal os. The endocervical canal may be filled up with mucus or blood. Embryos trapped in the mucus or blood after the passage of the endocervical canal may not be able to implant into the endometrium. Guardia™ Pro Protective ET catheter is designed to allow the safe passage of embryos through cervical mucus and blood as its outer sheath protects the embryo through entry and then opens in petals to further advance the inner catheter and gently place the embryo.

There is still no study comparing conventional and protective ET catheters in terms of the pregnancy rate of IVF treatment. The hypothesis of this study is that the pregnancy rate is significantly higher after ET using protective ET catheters.

Research plan Patients attending the Department for IVF-ET will be recruited if they fulfill the inclusion criteria and do not have the exclusion criteria. The FET treatment will be arranged as indicated.

On the day of ET, patients will be randomized according to a computer-generated randomization list in sealed envelopes into two groups: conventional and protective ET catheter groups. Conventional ET catheters will be used in the conventional ET catheter group while protective ET catheters will be used in the protective ET catheter group. Patients would be blinded to the group assigned although the clinical, nursing and laboratory staff will be aware of the type of catheters used.

A maximum of two good quality embryos are to be replaced. Patients are asked to keep a mildly full bladder so that the uterus can be visualized by abdominal sonogram during the procedure. A bivalve speculum is inserted into the vagina and the cervix is cleaned with warm saline and culture medium. The axis, degree of flexion and the configuration of the uterine cavity are determined by transabdominal ultrasound examination before the transfer. Under transabdominal ultrasound guidance, the outer catheter is inserted into the cervical canal 4 cm from the external os, with the tip just beyond the internal os. A malleable obturator is used if difficulty is encountered. The inner transfer catheter with the loaded embryo(s) is then inserted into the uterine cavity via the outer cannula. The aim is to put the tip of the inner catheter inside the uterine cavity 6 cm from the external os and care was taken not to advance the tip beyond 1 cm from the uterine fundus. The transfer volume is gently expelled by the technician. The catheters will be held in place for 30 seconds. Both the inner and outer catheters will be checked by the technician under the microscope to make sure that the embryos have been replaced.

The luteal phase support will be used if needed and antenatal management is as usual, if pregnant.

Sample size estimation The ongoing pregnancy rate of IVF-ET in 2010 was about 30.0%. Assuming a 10% increase following use of protective ET catheters as significant, 356 patients in each arm was required at a power of 80% and a significance level of 5% (Sigmastat, Jandel Scientific, San Rafael, CA, USA). A total of 720 patients will be recruited into the study.

Interim analysis will be performed after recruitment of every 100 subjects.

ELIGIBILITY:
Inclusion Criteria:

(i) ET in the fresh cycle (ii) Age <43 year (iii) Normal uterine cavity shown on ultrasound scanning

Exclusion Criteria:

(i) Three previous IVF cycles (ii) Natural IVF or IVM cycles (iii) Presence of hydrosalpinx on pelvic scanning (iv) Transfer of grade 5 embryos (v) Blastocyst transfer (vi) Use of donor oocytes (vii) Pre-implantation genetic diagnosis and (viii) Previously joined in the same study

Max Age: 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 10 weeks of gestation
  Pelvic ultrasound showed intrauterine pregnancy with fetal pulsation

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 weeks of gestation
  Pelvic ultrasound should an intrauterine sac with crown rump length corresponding to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China